CLINICAL TRIAL: NCT02725008
Title: A Randomized Double Blinded Placebo Controlled Trial of One Versus Two Doses of Oral Dexamethasone for the Treatment of Acute Asthma Exacerbation in the Pediatric Emergency Department (ED)
Brief Title: Trial of One Versus Two Doses of Dexamethasone for Pediatric Asthma Exacerbation
Acronym: R2D2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geoffrey W Jara-Almonte (Other)
Responsible Party: Sponsor-Investigator, Geoffrey W Jara-Almonte, Sub-Investigator, New York Presbyterian Brooklyn Methodist Hospital
Organization: New York Presbyterian Brooklyn Methodist Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 714220-1
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: Asthma; Pediatric; Emergency Department; Dexamethasone; Steroid
MeSH Terms: conditions — Asthma; Emergencies | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Patients are given one dose of oral dexamethasone 0.6 milligrams per kilogram up to 16 milligrams in the ED and a second dose of 0.6 milligrams per kilogram up to 16 milligrams to take 24 hours after ED visit
  Interventions: Drug: Dexamethasone
- Investigational (Experimental): Patients are given one dose of oral dexamethasone 0.6 milligrams per kilogram up to 16 milligrams in the ED and placebo to be taken 24 hours after ED visit
  Interventions: Drug: Dexamethasone; Drug: placebo

INTERVENTIONS:
Drug: Dexamethasone
  Other Names: decadron
Drug: placebo — to be given to the experimental group on the day after discharge from the ED in lieu of the second dose of dexamethasone
  Arms: Investigational

SUMMARY:
Comparing one versus two doses of oral dexamethasone for the treatment of asthma in the pediatric emergency department.

DETAILED DESCRIPTION:
A randomized double blinded placebo controlled trial comparing one dose of dexamethasone administered in the Emergency Department with two doses, the first given in the emergency department and the second 24 hours after the index ED visit.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma defined as at least two (2) prior episodes of respiratory illness characterized by wheezing treated with inhaled beta agonists

Exclusion Criteria:

* pregnancy
* severe chronic cardiac, respiratory, neurological or neuromuscular disease
* complete resolution of symptoms after one treatment of beta agonists
* severe asthma symptoms as defined by a Pulmonary Index Score of 12 or greater

Ages: 18 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelly, MD, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric Emergency Department
Pre-assignment Details: 99 participants were enrolled, 2 participants underwent initial enrollment but were not randomized to a group, leaving 97 participants who were assigned to a study group.
Groups:
- Control: Patients are given one dose of oral dexamethasone 0.6 milligrams per kilogram up to 16 milligrams in the ED and a second dose of 0.6 milligrams per kilogram up to 16 milligrams to take 24 hours after ED visit
  Dexamethasone
- Investigational: Patients are given one dose of oral dexamethasone 0.6 milligrams per kilogram up to 16 milligrams in the ED and placebo to be taken 24 hours after ED visit
  Dexamethasone
  placebo: to be given to the experimental group on the day after discharge from the ED in lieu of the second dose of dexamethasone
Period: Overall Study
Arm/Group | Control | Investigational
Started | 46 | 51
Completed | 37 | 39
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 7 | 9
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Admitted to hospital | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Investigational | Total
Number analyzed (Participants) | 46 | 51 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (6.0) | 7 (5.4) | 8.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 34 | 32 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 31 | 55
  White | 19 | 15 | 34
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 46 | 51 | 97
PIS Score [Median (Standard Deviation); unit: units on a scale] — Pulmonary Index Score - a clinical tool to assess severity of asthma exacerbation in children. Includes respiratory rate, amount of wheezing, I:E ratio, degree of accessory muscle use and oxygen saturation. Each subsection may be scored 0-3. Total score is arrived bu summation of sub-scores. Score range 0-15. Lower score corresponds to milder disease. <7 is considered mild, 7-12 moderate. Responsiveness to ED therapy (assessed by PIS Score at End of ED Stay) is expected to be an independent risk factor for the primary outcome, therefore it is considered a Baseline Measure.
  units on a scale
    PIS Score at ED arrival | 4 (2) | 5 (2.85) | 4 (2.53)
    PIS Score at End of ED Stay | 2 (1.35) | 1 (1.09) | 1 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: number of patients who experience any of the following outcomes - unplanned hospital admission for asthma symptoms, unplanned ED visit for asthma symptoms, unplanned urgent care visit for asthma symptoms, unplanned primary care physician visit for asthma symptoms, or prescription of a course of steroids
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Investigational
Number analyzed (Participants) | 37 | 39
Participants | 6 | 3
Statistical Analysis 1: Comparison: Control vs Investigational; Test type: Superiority; p = 0.3, Chi-squared; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.54 to 10.07]

2. Secondary Outcome: Change in Symptom Severity From Day 1 to Day 5
Description: Severity of asthma symptoms as reported by the Patient Self Assessment Score. Patients assessed severity of asthma symptoms in 4 categories (wheezing, coughing, activity and sleep) once per day during the 5 days between study enrollment and follow-up. Score range is 0 - 12 with 0 being mildest symptoms and 12 being most severe symptoms. Reported as change in score between enrollment (day 1) and follow-up (day 5).
Time Frame: 5 days
Population: Participants who had complete data available for analysis
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 22 | 11
score on a scale | -4 (3.39) | -4 (3.29)
Statistical Analysis 1: Comparison: Control vs Investigational; Test type: Superiority; p = 0.95, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Duration of study participation - 5 days
Arm/Group | Control | Investigational
All-Cause Mortality (participants affected / at risk) | 0/46 | 1/51
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/51
Other Adverse Events (participants affected / at risk) | 1/46 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=46) | Investigational (N=51)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=46) | Investigational (N=51)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Target enrollment was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02725008/Prot_SAP_000.pdf